CLINICAL TRIAL: NCT04242758
Title: Exploring the Association Between Phthalates Exposure, Measured Through Their Urinary Metabolites, and Renal Function Impairment in Individuals With TYpe 2 Diabetes - SGLT2 Subprotocol
Brief Title: Phthalates Exposure in Type 2 Diabetic Patients and Diuretic Therapy
Acronym: PURITY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Anna Solini, Associate Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PURITY - Protcol 5
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Renal Function Disorder; Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — dapagliflozin; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapaglifozin (Experimental): People undergoing SGLT2i (Dapaglifozin) therapy
  Interventions: Drug: Dapagliflozin 10 MG
- Hydrochlorothiazide (Experimental): People undergoing thiazide (Hydrochlorothiazide) therapy
  Interventions: Drug: Hydrochlorothiazide 12.5mg

INTERVENTIONS:
Drug: Dapagliflozin 10 MG — SGLT2-inhibitor: Diabetic oral drug with diuretic properties
  Other Names: DAPA
  Arms: Dapaglifozin
Drug: Hydrochlorothiazide 12.5mg — Best known thiazide class diuretic.
  Other Names: HCT
  Arms: Hydrochlorothiazide

SUMMARY:
In this open clinical trial, 30 subjects with inadequately controlled T2D and eligible, as per good clinical practice, for therapy with SGLT-2 inhibitor, will be randomized to receive a SGLT-2 inhibitor vs other oral-antidiabetic drugs (OADs) therapy for 3 months. Measures will be performed at baseline, after 2 days, after one month and at the end of the study protocol, as per good clinical practice

DETAILED DESCRIPTION:
* Total concentrations of MEHP, MEOHP and MEHHP will be quantified, in the laboratories of the Institute of Clinical Physiology, National Research Council, Pisa, in a spot morning urine sample by ultra-HPLC coupled with electrospray ionization/quadrupole time-of-flight mass spectrometry (Agilent UHPLC 1290 infinity coupled to an Agilent 6540 MS-QTOF, Santa Clara, CA) using stable isotope labeled substrates, i.e. MEHP (ring-1,2-13C2, dicarboxyl-13C2), MEHHP, MEHHP 13C4, MEOHP and MEOHP 13C4 that will be purchased from Cambridge Isotope Laboratories (Tewksbury, MA).
* Urinary creatinine concentrations will be measured to adjust urinary concentrations of DEHP metabolite (Beckman Coulter AU400, Brea, CA), thus minimizing the inﬂuence of urine volume.
* Serum and urinary inflammatory markers and adipocytokines will be quantitatively determined using sandwich enzyme-linked immunosorbent assays kits according to the manufacturer's instructions. Optical density will be measured using a microplate reader.
* Serum and urinary markers of oxidative stress will be measured by gold standard techniques. In detail, MDA will be quantified by TBARS reactive substances measured by optical density; GSH-Px by a specific assay kit according to the manufacturer's instruction; SOD activity will be determined using a specific SOD kit; urinary 8-isoprostane concentration will be measured by a specific affinity sorbent. (Cayman Chemical, Ann Harbor, MI, USA) according to the manufacturer's instructions.
* To analyze mitochondrial DNA we will apply a triplex design previously reported to amplify mitochondria loci located within the MinorArc and MajorArc, respectively. To assess nuclear DNA, we will use RNase P Copy Number Reference.
* The phthalates-free diet will be self-administered by the individuals under intervention, following a set of instruction and rules provided by the physicians based on the current literature data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sex;
* Age between 18 and 85 years;
* T2D
* T2D duration > 6 months
* BMI ≤ 40 Kg/m2,
* HbA1c > 48 mmol/mol
* Eligible for SGLT-2i therapy

Exclusion criteria

* age >85 years,
* eGFR <60 ml/min/1.73 m2,
* occurring acute complications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Urinary Phthalates concentration | Changes between baseline and 1 month
  Exposure to phthalates assessed through urinary concentration of phthalates metabolites spot and 24-hours
Urinary Phthalates concentration | Changes between baseline and 3 month
  Exposure to phthalates assessed through urinary excretion spot and 24-hours

SECONDARY OUTCOMES:
Fasting glucose | 1 and 3 months
  Fasting glucose measured in a fasting morning blood sample
Glycated Haemoglobin | 1 and 3 months
  HbA1c in a fasting measured in a morning blood sample
Renal function | 1 and 3 months
  Using creatinine measured in a fasting morning blood sample and estimated by eGFR (calculated with the CDK-EPI formula)
Macrovascular events | 1 and 3 months
  Number of participants with MACE events (Stroke, Acute Myocardial Infarction, Unstable Angina, Revascularization)
Albumin excretion | 1 and 3 months
  Measured by urinary albumin/creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Anna Solini, Prof, Principal Investigator — University of Pisa
Locations (1):
- University of Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dales RE, Kauri LM, Cakmak S. The associations between phthalate exposure and insulin resistance, beta-cell function and blood glucose control in a population-based sample. Sci Total Environ. 2018 Jan 15;612:1287-1292. doi: 10.1016/j.scitotenv.2017.09.009. Epub 2017 Sep 8. PMID 28898934
- [Background] Lind PM, Zethelius B, Lind L. Circulating levels of phthalate metabolites are associated with prevalent diabetes in the elderly. Diabetes Care. 2012 Jul;35(7):1519-24. doi: 10.2337/dc11-2396. Epub 2012 Apr 12. PMID 22498808
- [Background] Mengozzi A, Carli F, Biancalana E, Della Latta V, Seghieri M, Gastaldelli A, Solini A. Phthalates Exposure as Determinant of Albuminuria in Subjects With Type 2 Diabetes: A Cross-Sectional Study. J Clin Endocrinol Metab. 2019 May 1;104(5):1491-1499. doi: 10.1210/jc.2018-01797. PMID 30462244
- [Background] Kato K, Silva MJ, Reidy JA, Hurtz D 3rd, Malek NA, Needham LL, Nakazawa H, Barr DB, Calafat AM. Mono(2-ethyl-5-hydroxyhexyl) phthalate and mono-(2-ethyl-5-oxohexyl) phthalate as biomarkers for human exposure assessment to di-(2-ethylhexyl) phthalate. Environ Health Perspect. 2004 Mar;112(3):327-30. doi: 10.1289/ehp.6663. PMID 14998748
- [Background] Hauser R, Meeker JD, Park S, Silva MJ, Calafat AM. Temporal variability of urinary phthalate metabolite levels in men of reproductive age. Environ Health Perspect. 2004 Dec;112(17):1734-40. doi: 10.1289/ehp.7212. PMID 15579421
- [Background] Zota AR, Singla V, Adamkiewicz G, Mitro SD, Dodson RE. Reducing chemical exposures at home: opportunities for action. J Epidemiol Community Health. 2017 Jul 29;71(9):937-40. doi: 10.1136/jech-2016-208676. Online ahead of print. PMID 28756396
- [Background] Frederiksen H, Nielsen O, Koch HM, Skakkebaek NE, Juul A, Jorgensen N, Andersson AM. Changes in urinary excretion of phthalates, phthalate substitutes, bisphenols and other polychlorinated and phenolic substances in young Danish men; 2009-2017. Int J Hyg Environ Health. 2020 Jan;223(1):93-105. doi: 10.1016/j.ijheh.2019.10.002. Epub 2019 Oct 25. PMID 31669154